CLINICAL TRIAL: NCT01666756
Title: A Phase I Open Label Study Investigating the Combination of KD018 and Sorafenib (Nexavar) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Chinese Herbal Formulation PHY906 and Sorafenib Tosylate in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11043; NCI-2012-01324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5P01CA154295-02 (NIH)
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Advanced Adult Hepatocellular Carcinoma; BCLC Stage B Adult Hepatocellular Carcinoma; BCLC Stage C Adult Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — PHY 906; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Chinese herbal formulation PHY906 and sorafenib) (Experimental): Patients receive Chinese herbal formulation PHY906 PO BID on days 1-4, 8-11, 15-18, 21-24 and sorafenib tosylate PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Chinese herbal formulation PHY906; Drug: sorafenib tosylate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Dietary Supplement: Chinese herbal formulation PHY906 — Given PO
  Other Names: PHY-906; KD018
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of Chinese herbal formulation PHY906 when given together with sorafenib tosylate in treating patients with advanced liver cancer. Biological therapies, such as Chinese herbal formulation PHY906, may interfere with the growth of tumor cells and slow the growth of tumors. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may also stop the growth of liver cancer by blocking blood flow to the tumor. Giving Chinese herbal formulation PHY906 together with sorafenib tosylate may work better in treating advanced liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety and tolerability of KD018 (Chinese herbal formulation PHY906) in combination with daily sorafenib (sorafenib tosylate) and to determine the maximum tolerated dose (MTD) of the combination of KD018 plus sorafenib to bring forward into phase 2.

SECONDARY OBJECTIVES:

I. To describe the efficacy of the combination of KD018 plus sorafenib at the explored dose-levels in terms of best overall response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.

II. To assess the safety and tolerability of the combination of KD018 plus sorafenib as measured by the rate and severity of adverse events (AEs).

III. To determine the steady state of sorafenib after KD018 exposure at pre-dose and 1 hour and 2 hours post-dose at the explored combination dose-levels using concentrations at pre-dose (Cmin) and at 1 hour (C1h) and 2 hours (C2h) post-dose.

TERTIARY OBJECTIVES:

I. To assess the effect of treatment on soluble markers of angiogenesis, fibroblast growth factor (FGF), vascular endothelial growth factor (VEGF), placental growth factor (PLGF), soluble vascular endothelial growth factor receptor 1 (sVEGFR1), sVEGFR2, apoptosis (i.e. M30 monoclonal antibody [M30] and M65) and on the insulin-like growth factor (IGF) axis including molecules such as IGF-binding protein 2 (IGFII).

II. To correlate the above soluble biomarker measurements with clinical endpoints.

III. To examine the correlation between the soluble biomarkers.

IV. To examine the predictive relationship of immunohistochemical tumor biomarkers at baseline, i.e. phosphorylated ribosomal protein S6 kinase (pS6), p-protein kinase B (pAKT), p-mitogen-activated protein kinase 1 (ERK), p-mitogen-activated protein kinase kinase (pMEK), hypoxia-inducible factor 2, alpha subunit (HIF2a), phosphatase and tensin homolog gene (PTEN), signal transducer and activator of transcription 3 (acute-phase response factor) (STAT3) and tumor protein p53 (p53), as well as of mutational status, i.e. p53, phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) and PTEN, with efficacy endpoints (time to progression [TTP]).

V. To determine if soluble apoptosis markers (M30/M65) correlate with proliferative markers at baseline (proliferation-related Ki-67 antigen [Ki67] and p53) in archival tumor samples.

VI. To examine the relationship of immunohistochemical and/or soluble biomarkers with subgroup classification namely, patients with hepatitis B virus (HBV), patients with hepatitis C virus (HCV) and patients with other etiologies.

VII. To explore potential biomarker differences within patient subgroups, namely, patients with HBV, patients with HCV and patients with other etiologies.

VIII. To determine the effect of KD018 on cytokine/chemokine levels including interleukin (IL)-2, IL-4, IL-5, IL-6, IL-10, monocyte chemotactic protein 1 (MCP-1), tumor necrosis factor (TNF)-alpha, interferon (IFN)-alpha, VEGF, FGF-basic (b), sargramostim (GM-CSF), filgrastim (G-CSF).

IX. To explore potential relationships between efficacy and Cmin of sorafenib after co-administration with KD018 and between occurrence of adverse events and C1h/C2h endpoints (efficacy, safety, pharmacokinetics [PK]).

OUTLINE: This is a phase I, dose-escalation study of Chinese herbal formulation PHY906.

Patients receive Chinese herbal formulation PHY906 orally (PO) twice daily (BID) on days 1-4, 8-11, 15-18, 21-24 and sorafenib tosylate PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to take oral drugs
* Diagnosis of advanced hepatocellular carcinoma (HCC) according to the American Association for the Study of Liver Diseases (AASLD) guidelines
* HCC stage B or C according to the Barcelona Clinic Liver Cancer (BCLC)
* Previous or current use of sorafenib allowed
* Measurable disease according to RECIST, i.e. at least one measurable lesion; this lesion should not have been previously treated with local therapy; a treated lesion may be used where these lesions are the only lesions available for evaluation and have shown definite progression since their last local treatment; local therapy must have been completed at least four weeks prior to baseline evaluation
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Cirrhotic status of current Child-Pugh class A and B with no encephalopathy and no ascites (ascites controlled by diuretics is also excluded in this study); Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period
* For patients with positive HBV-deoxyribonucleic acid (DNA) and/or positive of hepatitis B surface antigen (HBsAg) results, they must be treated with anti-virals, as prophylaxis at least 1-2 weeks prior to receiving study drug, cycle 1, day 1
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 75000 x 10^6/L
* Hemoglobin (Hgb) >= 9 g/dL
* Alanine aminotransferase (ALT) =< 5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 x ULN
* Ability to understand and willingness to sign a written informed consent and to be able to follow the visit schedule
* Life expectancy of approximately 6 months
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for three months following duration of study participation; should a woman become pregnant, or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Previous or current use of sorafenib and previous use of tamoxifen is allowed as previous systemic therapy

Exclusion Criteria:

* Patients currently receiving any anti-cancer therapy, except sorafenib, or who have received any local anti-cancer therapy =< 4 weeks prior to baseline computed tomography (CT)/magnetic resonance imaging (MRI) scan, prior to cycle 1 treatment
* Active bleeding during the last 30 days prior to cycle 1 treatment including variceal bleeding (esophageal varices should be treated according to standard practice e.g. ligation/banding and procedure completed 30 days prior to cycle 1 treatment)
* Patients with a known hypersensitivity to KD018 or known hypersensitivity to sorafenib or contraindications to sorafenib based on the local sorafenib label
* Known history of human immunodeficiency virus (HIV) seropositivity (HIV testing is not mandatory)
* Any severe and/or uncontrolled medical conditions including:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction =< 6 months prior to cycle 1 treatment, serious uncontrolled cardiac arrhythmia, uncontrolled hypertension
  * Previous transient ischemic attack (TIA), cerebral vascular accident (CVA), symptomatic posterior vitreous detachment (PVD) within last 6 months of cycle 1 treatment
  * Congenital long QT syndrome
  * Patients with active alcohol intake
  * Acute and chronic, active infectious disorders and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy, in the opinion of the investigator, except chronic HBV or HCV
  * Impairment of gastrointestinal function or who have gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Patients receiving chronic treatment with corticosteroids (except for intermittent topical or local injection or aldosterone) or another immunosuppressive agent
* Patients treated with drugs known to be strong inhibitors or inducers of isoenzyme cytochrome P450, family 3, subfamily A (CYP3A) unless the drugs are medically necessary and no substitutes are available
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from surgery
* Patients who have received an investigative drug or therapy within the last 30 days prior to cycle 1 treatment
* Pregnant and/or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-06-11 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose, determined according to incidence of dose-limiting toxicity (DLT) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | 28 days

SECONDARY OUTCOMES:
Adverse events as determined by NCI CTCAE version 4 | Up to 4 weeks after completion of study treatment
Serious adverse events as determined by NCI CTCAE version 4 | Up to 4 weeks after completion of study treatment
Discontinuation rate | Up to 6 years
Dose adjustment rate | Up to 6 years
Tumor response in terms of best overall response, assessed using RECIST | Up to 6 years
Sorafenib tosylate concentration after co-administration with Chinese herbal formulation PHY906 | Baseline; 1 hour post-dose; 2 hours post-dose

OTHER OUTCOMES:
Change in cytokine/chemokine levels | Baseline to up to 6 years
Change in levels of soluble biomarkers | Baseline to up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chao, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States